CLINICAL TRIAL: NCT04082013
Title: Effect of Opposite Leg Position on Hamstring Flexibility in Patients With Mechanical Low Back Pain
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nasr Awad Abdelkader Othman, Lecturer of physical therapy for musculoskeletal Disorders, Cairo University
Other Study IDs: P.T.REC/012/002301
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2019-03

CONDITIONS: Flexibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hamstring Flexibility — The active knee extension test has been proposed as the gold standard for assessment of hamstring flexibility, as it utilizes readily available equipment and offers a quick, reliable, and low-cost alternative for measurement of hamstring flexibility (Connor et al; 2015).
  * The subject will be instructed to maintain 90° hip flexion in the supine position.
  * Then asked to actively extend the knee joint.
  * The degree of achieving active knee extension will be measured using a universal goniometer.
  * The average of three active knee extension measurements will be used as the hamstring muscle length for the data analysis (Dong-Kyu Lee, et al; 2018).
    * the procedures will be done with opposite-leg flexed, then repeated with opposite-leg extended.

SUMMARY:
PURPOSE: this study aimed to investigate the effect of opposite knee position on hamstring flexibility BACKGROUND Hamstrings tightness is one of the most common findings in patients with LBP. It is thought that, due to the attachments of hamstrings to the ischial tuberosity, hamstrings tightness generates posterior pelvic tilt and decreases lumbar lordosis, which can result in LBP.

HYPOTHESES There will be significant difference in the hamstring flexibility with changing position of opposite knee (flexed or extended) in patients with mechanical low back pain.

RESEARCH QUESTION: Will changing position of opposite knee (flexed or extended) affect the hamstring flexibility in patients with mechanical low back pain?

DETAILED DESCRIPTION:
* The subject will be instructed to maintain 90° hip flexion in the supine position.
* Then asked to actively extend the knee joint.
* The degree of achieving active knee extension will be measured using a universal goniometer.
* The average of three active knee extension measurements will be recorded used as the hamstring muscle length for the data analysis (Dong-Kyu Lee, et al., 2018).
* This test will be done for the same limb with opposite leg extended and with opposite flexed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of back pain and assessed with Mechanical inflammatory low back pain index and have very high grade for mechanical component.
* Age ranges from 18-40 years.
* The body mass index of the subject is ≤25 kg/meter square.

Exclusion Criteria:

1. Previous trauma, fractures or surgery of the back.
2. Malignancy of the back.
3. Rheumatoid arthritis
4. Spondylolysis or spondylolithesis
5. History of lower extremity injury within 6 months prior to the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Male and female
  * Age range from 18-40 years old
  * With previous mentioned inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Knee extension ROM | 30 minutes
  measuring knee extension ROM from 90 degrees hip flexion with opposite-leg flexed and extended

CONTACTS AND LOCATIONS:
Overall Officials: Nasr A. Abdelkader, PhD, Principal Investigator — Lecturer,Cairo University
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No